CLINICAL TRIAL: NCT06802510
Title: The Safety and Efficacy of Combined Microwave Ablation During Limb-sparing Surgery in High-risk Soft Tissue Sarcoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yu Zhang, PhD, Professor, Guangdong Provincial People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MWASTS001
Record Dates: First submitted 2025-01-21; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Sarcoma; Microwave; Ablation Techniques
Keywords: sarcoma; microwave ablation; limb-sparing surgery
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: Retrospective controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MWA group (Experimental): The MWA group received surgical resection combined with local lesion inactivation by MWA
  Interventions: Procedure: Microwave Ablation
- Control group (No Intervention): The control group received standard surgical resection.

INTERVENTIONS:
Procedure: Microwave Ablation — The MWA group followed a similar resection procedure as the control group. The area of ablation was evaluated strictly by radiologists and surgeons according to the following criteria: 1) Areas of tumor response, progression, or suspicious invasion (intermediate-high signal and edema range in T2) were assessed. Wide margins of at least 2-3 cm or more were obtained over the normal tissue around the tumor. Ablation margins were covered using a microwave ablation array with antennas (Microwave Ablation System BD-GT, Baird Medical LLC), aimed at completely inactivating the tumor in situ. Ablation needles were strategically arranged to form a matrix covering the target zone. The ablation time and power were determined based on the extent of the lesion, ensuring the temperature of the ablation area remained between 70-80°C. A 50 ml syringe was used to continuously drip and spray ice-cold saline to keep surrounding tissue temperatures below 40-43°C.
  Arms: MWA group

SUMMARY:
Soft tissue sarcoma (STS) is a rare, aggressive malignancy with a high risk of recurrence when invading surrounding structures, and the optimal treatment strategy for safe surgical margin is still unclear. This study aimed to evaluate the safety and efficacy of combined local inactivation by ablation in STS during limb-sparing surgery in high-risk STS patients.

DETAILED DESCRIPTION:
Soft tissue sarcoma (STS) is a rare, aggressive malignancy with a high risk of recurrence when invading surrounding structures, and the optimal treatment strategy for safe surgical margin is still unclear. This study aimed to evaluate the safety and efficacy of combined local inactivation by ablation in STS during limb-sparing surgery in high-risk STS patients. Investigators collected data retrospectively from participants diagnosed with soft tissue sarcoma who were treated at a tertiary medical institution from January 1, 2018, to December 31, 2022. This study was approved by the hospital's Ethics Committee (XJS2022-101-01), and all participants provided written informed consent. The participants were divided into two groups (MWA and control group). The MWA group received surgical resection combined with local lesion inactivation by MWA, while the control group underwent standard surgical resection alone. Non-specified sarcomas are treated with the AI(Doxorubicin+Ifosfamide) chemotherapy regimen, while Ewing's sarcoma is treated with the standard recommended VDC ((Vincristine + Doxorubicin + Cyclophosphamide)/IE(Ifosfamide + Etoposide) chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed soft tissue sarcoma (FNCLCC grade G2-G3);
2. MRI/CT confirmed tumor invasion beyond anatomical compartments, joint involvement, or encroachment on surrounding tissues (bones, muscle, etc.);
3. After being fully informed of the risks, the patient strongly refuses amputation or wide resection, which leads to irreversible impaired function.
4. Good physical condition, able to tolerate surgery;

Exclusion Criteria:

1. Patients with distant metastasis at the time of initial diagnosis;
2. Patients with missing clinical or follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-01-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of diagnosis until the date of documented death, assessed up to 5 years (up to 5 year)
  Overall survival was defined as the time from diagnosis to last follow-up or death.
progression-free survival (PFS) | From date of surgery until the date of first documented disease progression or death, assessed up to 5 years
  progression-free survival (PFS) was the time from surgery to disease progression or death
Local disease-free survival (DFS) | From date of surgery until the date of first documented local tumor recurrence, assessed up to 5 years
  Local disease-free survival (DFS) was the time for local tumor recurrence after surgery.

SECONDARY OUTCOMES:
Postoperative complications | Post-operation 3 months
  Serious postoperative complications were recorded according to CTCAE 4.0, including severe wound healing problems, deep infections, bone necrosis, wound burn, persistent pain, and major neurovascular injuries.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong provincial people's hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Due to ethical and patient privacy restrictions, relevant data is not publicly disclosed